CLINICAL TRIAL: NCT01908036
Title: Use of a Monitor in ME/CFS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York CFS Association (Other)
Responsible Party: Sponsor
Other Study IDs: FITBIT2
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic fatigue syndrome; CFS; myalgic encephalomyelitis; M.E.; activity monitor
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The use of an activity monitor to determine increase or decrease of activity in patients suffering from chronic fatigue syndrome.

DETAILED DESCRIPTION:
A cohort of 50 patients suffering from chronic fatigue syndrome will be given an informed release form. Have a signed the informed release they will be given a Fitbit activity monitor. These monitors will be evaluated on a weekly interval by computer interface. The activity will be calculated to determine the online of activity and whether there is increase or decrease in activity during the time of the study. The study is an observational rather than an interventional study. There is no invasion or intervention in the patient's normal activities

ELIGIBILITY:
Inclusion Criteria:

Fukuda and Canadian consensus criteria for the diagnosis of chronic fatigue syndrome

Exclusion Criteria:

Acute disease and exclusion conditions in Fukuda criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 CFS patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
observation of activity level in CFS patients | 6 months
  observation of activity level in CFS patients using objective activity monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Me/Cfs Center,860 Fifth Avenue, New York, New York, United States